CLINICAL TRIAL: NCT04185259
Title: Efficacy of Acupuncture vs Sham Acupuncture or Waitlist Control for Patients With Chronic Planter Fasciitis: Study Protocol for a 2-center Randomized Controlled Trial
Brief Title: Acupuncture vs Sham Acupuncture or Waitlist Control for Patients With Chronic Planter Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, weiming wang, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZZ13-YQ-019
Record Dates: First submitted 2019-11-30; First posted 2019-12-04 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to acupuncture group, sham acupuncture group, or waitlist (no acupuncture) group at a ratio of 2:1:1 using simple randomization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants in acupuncture group and sham acupuncture group, together with efficacy evaluators and data analysts will be blinded to the group assignments. Participants in the waitlist control group and acupuncturists will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture group (Experimental)
  Interventions: Other: Acupuncture
- Sham acupuncture (Sham Comparator)
  Interventions: Other: Sham acupuncture
- Waitlist control group (No Intervention): Participants will receive no treatment for their heel pain for a period of 16 weeks after randomization, and subsequently have the option of 4 weeks (12 sessions) of acupuncture with free of charge at the end of follow-up.

INTERVENTIONS:
Other: Acupuncture — The investigators will apply two Ashi points (the two most severe tender points in the most sensitive area over the anteromedial aspect of the heels), Chengshan (BL57), Taixi (KI3) and Kunlun (BL60) in this trial. With the patient in a prone position, the local skin will be routinely sterilized followed by a 10mm diameter and 5mm thick sterile adhesive pad pasting onto each selected acupoint. Ashi points will be perpendicularly inserted through the pad to the plantar fascia layer with a depth of approximately 15-20mm depending on the location. BL57, KI3 and BL60 will be punched perpendicularly 10-15mm deep into the skin through the pad. All needles except Ashi points will be manually stimulated by small, equal manipulations of lifting, thrusting, twirling and rotating to achieve De qi. Needles will be retained for 30 minutes per treatment. During each treatment, every needle will be manipulated three times every 10 minutes.
  Arms: Acupuncture group
Other: Sham acupuncture — Sham Ashi (0.5 cun away from Ashi, one 'cun' is equivalent to the greatest width of the individual patients' thumb, ~1.5 cm), sham BL57 (0.5 cun lateral to true BL57 horizontally), sham KI3 (midway between true KI3 and heel tendon) and sham BL60 (midway between true BL60 and heel tendon) will be used. Treatment protocol will be similar to that of the acupuncture group. The Hwato-brand disposable blunt-tipped needles (size 0.30 × 25 mm) will be inserted at sham points through adhesive pads to the skin without skin penetration. The needles will then be lifted, thrusted, twirled, and rotated evenly three times every ten minutes. No specific de qi response will be elicited.
  Arms: Sham acupuncture

SUMMARY:
Plantar fasciitis (PF) predominantly affects elderly and middle-aged individuals and is more frequent in runners or those whose employment requires standing. The available treatment options of PF mainly included non-operative treatments (e.g., plantar fascia and gastrocnemiussoleus muscle stretching, heel cups, arch supports, night splints, nonsteroidal antiinflammatory drugs (NSAIDs), local corticosteroid injections) and operative management. However, no consensus has been reached regarding the most beneficial treatment method for PF.

Acupuncture has been used in the management of PF and the other musculoskeletal pain-related conditions for thousands of years. Recent two systematic reviews have found that acupuncture may reduce pain intensity and improve plantar function for patients with PF. However, there are methodological problems with small sample size, or not controlled with a placebo/waitlist group, or not account for the confounding effects of patients who experienced combination treatments in the design of the included acupuncture literature. Therefore, the placebo effect of acupuncture and a possible spontaneous remission for PF cannot be excluded and the beneficial effects of acupuncture for PF remained need to more assessment.

The investigators designed a randomized controlled trial to evaluate the efficacy of Traditional Chinese acupuncture (TCA), compared with sham acupuncture (SA) or being on a waitlist control group (no acupuncture treatment), for patients with chronic PF for ≥ 6 months. The hypothesis was that combined acupuncture and sham acupuncture will result in larger improvements in heel pain more than no acupuncture treatment in patients with chronic PF. Secondary hypotheses examined whether acupuncture reduce heel pain intensity more effectively than sham acupuncture or no acupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years;
2. History of planter medial heel pain for at least 6 months before enrolment;
3. Reported an average worst pain intensity at first steps in the morning over the last 7 days of at least 50mm on a 100-mm visual analog scale (VAS) before enrolment;
4. Failure to respond to conservative treatment for ≥ 1 months, including any of the following modalities: stretching exercises, nonsteroidal anti-inflammatory drugs, orthotics;
5. Ability to comply with the study protocol, understand the medical information forms as well as having signed informed consent.

Exclusion Criteria:

1. History of calcaneus fracture, calcaneal bone tumor or cyst, plantar fascia rupture， or have a significant foot deformity(clubfoot, pes cavus, or pes calcaneovalgus);
2. Previous injection (corticosteroid, platelet-rich plasma, lidocaine needling), or radiation, or surgery to plantar fascia within 6 months preceding enrollment;
3. Radiculopathy or peripheral neuropathy around the ankle joint such as nerve entrapment tarsal tunnel syndrome or Achilles tendinopathy;
4. Systemic disorders like rheumatoid arthritis, gout, Reiter syndrome, type 1 or 2 diabetes mellitus, osteoporosis, spondyloarthritis, or osteomyelitis;
5. Joint, bone, or skin infection in the affected foot;
6. Clinically significant cardiovascular disorder, severe hepatic/renal insufficiency or coagulation disorder at baseline as determined by the investigator;
7. Known phobic to acupuncture or received acupuncture treatment within 4 weeks prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with treatment response 4 weeks after randomization | at week 4
  A treatment responder is defined as a participant having a minimum of 50% improvement in the worst pain intensity during the first steps in the morning compared with baseline.

SECONDARY OUTCOMES:
Changes in VAS score for worst pain intensity during the first steps in the morning from baseline to 4 weeks, 8 weeks and 16 weeks after randomization | at week 4, week 8 and week 16
  Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain.
Changes in VAS score for mean pain intensity during the day from baseline to 4 weeks, 8 weeks and 16 weeks after randomization | at week 4, week 8 and week 16
  Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain.
Changes in the pressure pain threshold (PPT) at the most painful area from baseline to 4 weeks, 8 weeks and 16 weeks after randomization | at week 4, week 8 and week 16
  Pressure pain threshold (PPT) is defined as the minimum pressure detected when the sensation of pressure changes to a first sensation of pain, PPT will be tested with a pressure algometer (Fabrication Enterprises, Inc., White Plains, NY; from 1 kg/cm2 to 5 kg/cm2) involved a metal probe with a 0.5 cm2 rubber disc by a trained researcher.
Changes in ankle range of motion (AROM) from baseline to 4 weeks, 8 weeks and 16 weeks after randomization | at week 4, week 8 and week 16
  The examiner will measure the AROM including plantar dorsiflexion and plantar flexion using a digital goniometer (Tangxia Electronic Instrument Factory, Dongguan, from 0° to 360°).
Changes in Foot and Ankle Ability Measure (FAAM) total score and subscale scores from baseline to 4 weeks, 8 weeks and 16 weeks after randomization | at week 4, week 8 and week 16
  The Foot and Ankle Ability Measure has a maximum potential score (116 total, 84 ADL, and 32 Sport subscales). The obtained score (total score, ADL, and sport subscale scores) is divided by the maximum potential score and multiplied by 100 to get a percentage.
Change in plantar fascia thickness (PFT) from baseline to 4 weeks after randomization | at week 4
  Plantar fascia thickness (PFT) will be measured at the thickest point closest to the calcaneal insertion in its medial portion using ultrasound
Participant global assessment of improvement | at week 4, week 8 and week 16
  Participants will be asked to rate his/her global improvement using a 7-point scale. The improvement will be scale from 1(complete recovery) to 7(vastly worse), with 2 being obvious improvement, 3 being a little improvement, 4 being no change, 5 being a little worse and 6 being obvious worse.
The proportion of patients using rescue medicine and the mean frequency of rescue medicine use per week during weeks 1-4 and weeks 5-16 | weeks 1-4, and weeks 5-16
  The proportion of patients using rescue medicine and the mean frequency of using rescue medicine per week will be compared among three groups during weeks 1-4, and weeks 5-16.

OTHER OUTCOMES:
Participants'expectation towards acupuncture | at baseline
  Participants in acupuncture group and sham acupuncture group will be asked that "Do you think acupuncture will be helpful to improve your chronic PF?" Participant will choose one of the following answers: "Extremely helpful", "Very helpful", "Helpful", "Not help at all" and "Unclear"
The proportion of participants who have maintained blinding during treatment in acupuncture and SA groups | at week 4
  Participants' blindness to the mode of acupuncture will be assessed five minutes after the end of any treatment in the fourth week by asking the patients the following question: "Which of the two acupuncture modalities that you have received, acupuncture or SA?" Participants will choose one of the following answers: "Acupuncture", "Sham acupuncture", or "Unclear"
Incidence of adverse events | weeks 1-16
  The adverse events (AEs) during the whole study will be recorded and described as acupuncture-related AEs and non-acupuncture-related AEs. Acupuncture-related AEs include fainting, broken needle, unbearable pain during acupuncture (VAS ≥ 8, using a 0[no pain] to10 [worst pain imaginable] VAS), and other unintended signs, or symptoms after acupuncture (e.g., localized haematoma or infection, nausea, dizziness, vomiting, headache, palpitations). Detailed information on AEs including the name, onset and end date, intensity, correlation with acupuncture and outcome will be detailed documented in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, MD, PhD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Department of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences Guang'anmen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang W, Liu S, Liu Y, Zang Z, Zhang W, Li L, Liu Z. Efficacy of acupuncture versus sham acupuncture or waitlist control for patients with chronic plantar fasciitis: study protocol for a two-centre randomised controlled trial. BMJ Open. 2020 Sep 25;10(9):e036773. doi: 10.1136/bmjopen-2020-036773. PMID 32978188